CLINICAL TRIAL: NCT00805584
Title: A Multi-center, Open-label, Non-comparative Study of the Relief of Nasal Symptoms and Tolerability in Subjects With Seasonal Allergic Rhinitis (SAR) Treated With Aerius.
Brief Title: Study of Nasal Symptom Relief and Side Effects in Hayfever Patients Treated With Aerius (Desloratadine)(P03442)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03442
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: desloratadine

INTERVENTIONS:
Drug: desloratadine — Aerius (desloratadine) tablets; 5mg orally once a day in the morning for 15 days
  Other Names: Aerius, Clarinex, SCH 34117, descarboethoxyloratadine

SUMMARY:
The purpose of this study was to test the effectiveness and side effects of desloratadine (Aerius) in patients with hayfever. Patients took desloratadine once a day for 15 days. At the end of therapy, they scored how severe their hayfever symptoms were and how they responded to therapy. Side effects were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >=18 years of age, of either sex and any race.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using or agree to use an acceptable method of birth control. Women who are not currently sexually active must agree and consent to use some sort of contraception should they become sexually active while participating in the study.
* Subjects must be in general good health, i.e., they must be free of any clinically significant disease (other than SAR) that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules, and agree to report concomitant medications and adverse events to the Investigator or designee.
* Subjects must have at least a positive history, self-reported history of signs and symptoms is acceptable, of recurring seasonal allergic rhinitis
* Subjects must be clinically symptomatic with SAR at Visit 2 (Baseline): the total (nasal + non-nasal) symptom score must be >=8 points with a nasal congestion score of >=2, and the non-nasal symptom score must be >=2. Subjects may be rescheduled up two additional times for the qualifying visit if they do not meet the minimum symptom scores.
* Women of childbearing potential must have be negative pregnancy history at Visit 1.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.
* Subjects with asthma who require chronic use of inhaled or systemic corticosteroids.
* Subjects with current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip.
* Subjects with rhinitis medicamentosa.
* Subjects who have had an upper respiratory tract or sinus infection that required antibiotic therapy within 14 days prior to Visit 1 (Screening / Consent), or subjects who have had a viral upper respiratory infection within 7 days prior to Visit 1.
* Subjects who have nasal structural abnormalities, including nasal polyps and marked septal deviation, that significantly interferes with nasal airflow.
* Subjects who, in the opinion of the Investigator, are dependent upon nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids.
* Subjects with a history of hypersensitivity to desloratadine or any of its excipients.
* Subjects who are staff personnel directly involved with the administration of this study.
* Subjects who have any current evidence of clinically significant hematopoetic, metabolic, cardiovascular, immunologic, neurologic, hematologic, gastrointestinal, hepatic, renal, psychiatric, cerebrovascular, or respiratory disease, or any other disorder which, in the judgment of the Investigator, may interfere with the study evaluations or affect subject safety.
* Subject taking prohibited drugs listed in the study protocol are excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2003-05; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Relief of allergy symptoms | Baseline and end of therapy

SECONDARY OUTCOMES:
Global therapeutic response | End of therapy
Adverse events | Baseline and end of therapy